CLINICAL TRIAL: NCT06193941
Title: Research on the Accurate Diagnosis of Urinary Tract Tumors and the Development of Kits
Status: Completed | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: W20231218
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Bladder Cancer; Urothelial Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Case group （bladder cancer）: Urine exosomes were enriched for RT-qPCR within 4 hours after samples were collected.
  Interventions: Diagnostic Test: RT-qPCR
- Control group （benigh）: Urine exosomes were enriched for RT-qPCR within 4 hours after samples were collected.
  Interventions: Diagnostic Test: RT-qPCR
- Healthy people group: Urine exosomes were enriched for RT-qPCR within 4 hours after samples were collected.
  Interventions: Diagnostic Test: RT-qPCR

INTERVENTIONS:
Diagnostic Test: RT-qPCR — RT-qPCR

SUMMARY:
Bladder cancer is the second most prevalent urological malignancy worldwide, with a high incidence and poor patient prognosis. Achieving early diagnosis and intervention for bladder cancer is one of the most important ways to improve clinical management and patient prognosis. Tumor exosomes can be released into biological fluids at an early stage of a tumor, and many studies have shown that exosomal RNA can be used as a reliable biomarker to diagnose tumors in a non-invasive way. Based on the clinical needs for early diagnosis of bladder cancer, we aim to screen several early diagnostic markers with potential predictive value, establish an early diagnostic model for bladder cancer, and validate the validity and reliability of this diagnostic model through a large-scale clinical cohort to complement the diagnosis of early-stage cancers and to improve the rate of early diagnosis of cancer.

DETAILED DESCRIPTION:
In response to the clinical demand for accurate early diagnosis of bladder cancer, this project aims to gradually conduct in-depth research on precise early diagnosis of bladder cancer. This includes establishing key techniques for efficient and convenient enrichment of exosomes, identifying potential exosome biomarkers for bladder cancer based on bladder cancer transcriptome sequencing data, and conducting large-scale clinical cohort studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years with defined gender;
2. Preoperative patients are preliminarily evaluated as bladder tumors by cystoscopy, FISH, cytology, or imaging.

Exclusion Criteria:

1. Aged <18 years;
2. Post-operative or after anti-tumor treatment such as chemotherapy or immunotherapy
3. History of other malignant tumors
4. Specimens with hemolytic conditions;
5. Patients with incomplete, undocumented, and uncooperative data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with bladder cancer treated in Zhongnan Hospital of Wuhan University
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
RT-qPCR | Urine exosomes were enriched for RT-qPCR within 4 hours after the samples were collected.
  Urine exosomal RNA

CONTACTS AND LOCATIONS:
Overall Officials: Fubing Wang, Doctor, Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China